CLINICAL TRIAL: NCT04498507
Title: Psychosocial Outcomes in Families of Patients Admitted in ICU for COVID-19 During the Pandemic in Belgium
Brief Title: Psychosocial Outcomes in Families of COVID-19 ICU Patients
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, MD, PhD, University of Liege
Other Study IDs: Family COVID
Record Dates: First submitted 2020-08-01; First posted 2020-08-04 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Critical Illness; Family; Psychological Stress; Covid19
MeSH Terms: conditions — Critical Illness; Stress, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HADS questionnaire — Patients will be asked to answer to 3 questionnaires about anxiety and depression, post-traumatic stress disorder and health-related quality of life
  Other Names: IES-R questionnaire; EQ-5D questionnaire

SUMMARY:
During the first part of the SRAS-COV2 pandemic, families were not allowed to visit the patients in ICU. We know that families can develop "Family-PICS" after their relatives' ICU stay. The aim of the study is to study the psychosocial outcomes of families of patients who were admitted in ICU for COVID-19 during the pandemic. The second objective was to search for any differences in outcomes whether families benefited from video-conferences with the medical team and their relatives or not during the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* the referent family member of any patient admitted in ICU for COVID-19 during the first part of the pandemic

Exclusion Criteria:

* cognitive disorders
* not French-speaking
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: this study includes the family members of patients who were admitted in ICU for sever COVID-19 during the first part of the pandemic when visits in ICU were not allowed
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
occurence of anxiety and depression | one month after ICU discharge
  sub scores of HADS questionnaire >7
occurence of anxiety and depression | three months after ICU discharge
  sub scores of HADS questionnaire >7
occurence of acute stress | one month after ICU discharge
  IES-R score > 22
occurence of post-traumatic stress disorder | three months after ICU discharge
  IES-R score > 36
quality of life | one month after ICU discharge
  assessed using the EQ-5D questionnaire
quality of life | three months after ICU discharge
  assessed using the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No